CLINICAL TRIAL: NCT06924879
Title: The Effects of the Mindfulness -Based Pregnancy Stress Reduction Program on the Stress Levels, Sleep Quality and Awareness Levels of Pregnant Women
Brief Title: The Effects of the Mindfulness-Based Pregnancy Stress Reduction Program on Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Gülendan Güntürk, Master's degree student, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2024-363
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Pregnancy
Keywords: pregnancy; stress; sleep quality; nursing; mindfulness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The study consists of two groups: experimental and control group. In the study, while the control group will receive routine pregnancy care, the experimental group will receive an 8-session mindfulness-based pregnancy stress reduction program.
  Before randomization, pregnant women who meet the inclusion criteria will be informed about the study, their verbal and written consent will be obtained for participation in the study, and then pretest data will be collected. Personal Information Form, Tilburg Distress in Pregnancy Scale, Pittsburgh Sleep Quality Index and Mindfulness Scale will be used to collect pretest data from pregnant women who agree to participate in the study. After the pre-test data are collected, the pregnant women will be randomly assigned to one of the intervention and control groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: In the study, in order to prevent selection bias, pregnant women randomly assigned to the intervention or control group by randomization method will not know which group they are in. However, since the researcher will know which group the pregnant women are in, one-way blinding will be performed during the data collection phase of the study. Since a statistical expert other than the researchers will perform the statistical analysis of the data obtained as a result of the research, two-way blinding will be performed at the statistical analysis stage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnant women participating in a mindfulness-based stress reduction program (Experimental): The Mindfulness-Based Pregnancy Stress Reduction Program consisting of 8 sessions will be applied to the pregnant women included in the intervention group and post-test data will be collected with measurement tools in the last trimester of pregnancy and 1-3 months after delivery after the training.
  Interventions: Other: Mindfulness-Based Pregnancy Stress Reduction Program
- Pregnant women not participating in a mindfulness-based stress reduction program (No Intervention): Pregnant women in the control group will not receive any intervention and will receive routine pregnancy care and practices. Post-test data will be collected from the pregnant women in the control group in the last trimester of pregnancy and between 1-3 months after delivery with measurement tools. After the post-test data are collected, the pregnant women in the control group will also receive mindfulness training.

INTERVENTIONS:
Other: Mindfulness-Based Pregnancy Stress Reduction Program — Mindfulness-Based Pregnancy Stress Reduction Program Training Content Session 1 Introduction to the program Course preparation Orientation process Session 2 Introduction to Mindfulness practices Session 3 Focusing on the moment Session 4 Coping with thoughts Connecting with pregnant women's bodies Becoming aware of their thoughts, feelings and bodily senses Session 5 Releasing emotions and thoughts Session 6 Awareness Session 7 Keeping distance from thoughts Session 8 Accepting Awareness
  Arms: Pregnant women participating in a mindfulness-based stress reduction program

SUMMARY:
This study was planned as a randomized controlled experimental study to determine the effect of Mindfulness-Based Pregnancy Stress Reduction Program on stress levels, sleep quality and mindfulness levels of pregnant women.

Hypotheses of the Study:

Hypothesis 1 (H1): Mindfulness-Based Pregnancy Stress Reduction Program has an effect on reducing stress levels of pregnant women.

Hypothesis 2 (H1): Mindfulness-Based Pregnancy Stress Reduction Program has an effect on improving sleep quality of pregnant women.

Hypothesis 3 (H1): Mindfulness-Based Pregnancy Stress Reduction Program has an effect on increasing the mindfulness levels of pregnant women.

Hypothesis 4 (H1): Mindfulness-Based Pregnancy Stress Reduction Program has an effect on reducing women's stress levels in the postpartum period.

Hypothesis 5 (H1): Mindfulness-Based Pregnancy Stress Reduction Program has an effect on improving women's sleep quality in the postpartum period.

Hypothesis 6 (H1): Mindfulness-Based Pregnancy Stress Reduction Program has an effect on increasing women's mindfulness levels in the postpartum period.

It is planned to collect the research data from pregnant women who applied to the obstetrics and gynecology outpatient clinics of Vezirköprü State Hospital by face-to-face interview technique using Personal Information Form, Tilburg Distress in Pregnancy Scale, Pittsburgh Sleep Quality Index, Perceived Stress Scale and Mindfulness Scale.

It is planned to collect the research data in three stages. In the first stage, pre-test data will be collected from all pregnant women in the intervention and control groups who applied to the obstetrics outpatient clinic of Vezirköprü State Hospital, met the inclusion criteria and agreed to participate in the study. Pregnant women in the intervention group will be applied the Mindfulness-Based Pregnancy Stress Reduction Program consisting of 8 sessions and post-test data will be collected with measurement tools in the last trimester of pregnancy and 1-3 months after delivery. Pregnant women in the control group will not receive any intervention and will receive routine pregnancy care and practices. Post-test data will be collected from the pregnant women in the control group in the last trimester of pregnancy and between 1-3 months postpartum with measurement tools. After the post-test data are collected, the pregnant women in the control group will also receive mindfulness training.

DETAILED DESCRIPTION:
This study was planned as a randomized controlled experimental study to determine the effect of Mindfulness-Based Pregnancy Stress Reduction Program on stress levels, sleep quality and mindfulness levels of pregnant women. This study have been conducted between June 01, 2024 and December 31, 2024 in the obstetrics outpatient clinics of Vezirköprü State Hospital affiliated to Samsun Provincial Health Directorate. There are two obstetrics outpatient clinics, breastfeeding counseling/lactation-relactation outpatient clinic and a pregnancy school in the hospital where the research will be conducted. In addition to the outpatient clinics, there are pregnancy monitoring and nonstress testing rooms.

The population of the study will consist of pregnant women who applied to the Obstetrics and Gynecology Outpatient Clinics of Vezirköprü District State Hospital affiliated to Samsun Provincial Health Directorate. Pregnant women who applied to Vezirköprü District State Hospital Obstetrics and Gynecology Outpatient Clinics and met the criteria for inclusion in the sample will be included in the sample of the study.

In order to determine a significant group effect in the sample calculation of the study, the minimum sample size was calculated as 33 pregnant women in the intervention group, 33 pregnant women in the control group, and 66 pregnant women in total, using an alpha margin of error of 0.05, a research power of 0.80 and an intermediate group effect (partial eta squared) of 0.03. In order to strengthen the results of the study and increase reliability and against the possibility of sample loss during the study, it was decided to include 80 pregnant women (40 intervention and 40 control), which is 20% more than the sample size.

It is planned to collect the research data from pregnant women who applied to the obstetrics and gynecology outpatient clinics of Vezirköprü State Hospital by face-to-face interview technique using Personal Information Form, Tilburg Distress in Pregnancy Scale, Pittsburgh Sleep Quality Index, Perceived Stress Scale and Mindfulness Scale.

It is planned to collect the research data in three stages. In the first stage, pre-test data will be collected from all pregnant women in the intervention and control groups who applied to the obstetrics outpatient clinic of Vezirköprü State Hospital, met the inclusion criteria and agreed to participate in the study. Pregnant women in the intervention group will be applied the Mindfulness-Based Pregnancy Stress Reduction Program consisting of 8 sessions and post-test data will be collected with measurement tools in the last trimester of pregnancy and 1-3 months after delivery. Pregnant women in the control group will not receive any intervention and will receive routine pregnancy care and practices. Post-test data will be collected from the pregnant women in the control group in the last trimester of pregnancy and between 1-3 months postpartum with measurement tools. After the post-test data are collected, the pregnant women in the control group will also receive mindfulness training.

ELIGIBILITY:
Inclusion Criteria:

* - Volunteering to participate in the research,
* Be over 18 years of age,
* Being literate,
* To be able to understand and speak Turkish,
* Nulliparous conception,
* Don't be a singleton,
* Gestational age between 24-32 weeks.

Exclusion Criteria:

* - Multiparous pregnancy,
* Don't have a high-risk pregnancy,
* Do not have a diagnosed psychiatric illness,
* Conception as a result of infertility treatment,
* Attending childbirth preparation courses
* Planning a cesarean birth
* Previous experience of yoga and meditation,
* Don't want to leave the research,
* Not attending any session of the Mindfulness-Based Pregnancy Stress Reduction Program
* Failure to complete the data collection tools completely.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study was administered to pregnant women.
Enrollment: 80 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Tilburg Distress Scale in Pregnancy | From participation until the end of the 8th week
  The Tilburg Distress Scale in Pregnancy was developed to determine distress in pregnancy. The scale, which can be applied to pregnant women twelve weeks and over, consists of 16 items and is graded on a 4-point Likert scale (very often 0 points, quite often 1 point, occasionally 2 points, rarely/never 3 points). The total score that can be obtained from the scale varies between 0 and 48. According to the cut-off point, a total score of 28 and above indicates that the pregnant woman is at risk for distress. Items numbered 3, 5, 6, 7, 9, 10, 10, 11, 12, 13, 14, 16 in the scale are reverse coded. The scale has 2 sub-dimensions, "negative affect" consisting of 11 items and "partner involvement" consisting of 5 items. The items numbered 1, 2, 4, 8 and 15 in the scale belong to the "spousal involvement" sub-dimension, while the other items belong to the "negative affect" sub-dimension.
Pittsburgh Sleep Quality Index | From participation until 1 to 3 months postpartum
  Pittsburgh Sleep Quality Index is a scale to assess sleep quality in psychiatry and clinical studies. The scale evaluates sleep disturbances and sleep quality in the last 1 month. The Turkish validity and reliability of the scale was performed by Agargün et al. Pittsburgh Sleep Quality Index consists of 24 questions and 7 sub-dimensions. These sub-dimensions are "subjective sleep quality", "sleep delay", "sleep duration", "habitual sleep efficiency", "sleep disturbance", "sleep medication use" and "daytime dysfunction". Each sub-dimension is evaluated with a score between 0-3 and the total scores of the sub-dimensions give the scale score. The total score of the scale is between 0-21. If the total score obtained from the scale is above 5, it is clinically evaluated as poor sleep quality (Agargün, 1996). Agargün et al. (1996) found the Cronbach's alpha reliability coefficient of the scale to be 0.804.
Perceived Stress Scale | until the 1st to 3rd months after birth
  The Perceived Stress Scale was developed to determine the extent to which individuals perceive certain situations in their lives as stressful. Its Turkish validity and reliability was conducted by Eskin et al. The Perceived Stress Scale consists of 10 items and measures how stressful people perceive some situations in their lives. The scale is a five-point Likert scale and is scored as 0 "never", 1 "almost never", 2 "sometimes", 3 "often", 4 "very often". The scores of the items containing 7 positive statements in the scale are reversed and the total score of the scale is obtained by adding the scores of the other items. Scores between 0-56 can be obtained from the scale. There is no cut-off point in the scale, and an increase in the score indicates that the stress perception of the individual is high. Eskin et al. (2013) found the Cronbach's alpha internal consistency coefficient of the scale to be 0.84.

SECONDARY OUTCOMES:
Mindfulness Scale | From participation until 1 to 3 months postpartum
  The Mindfulness Scale (MBAS), developed to measures individual differences in attention and awareness skills towards momentary experiences (Brown & Ryan, 2003).The Mindfulness Scale aims to determine whether there is awareness and attention in relation to what is happening in the present rather than elements related to mindfulness such as acceptance, trust, and co-sensation. It is used to assess individual differences in the frequency of mindfulness. It consists of 15 items, each with declarative and affirmative statements. The Mindfulness Scale measures how often individuals experience a particular situation using a 6-point Likert scale. Scores are between 1 and 6. The lowest score that can be obtained from the scale is 15 and the highest score is 90. A high score on the scale means that the level of mindfulness is high. Özyeşil et al. (2013) calculated the internal consistency coefficient of the scale as 0.82 and the test-retest correlation as 0.86.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Akman, PhD lecturer, Study Director — Ondokuz Mayıs University
Locations (1):
- Vezirkopru County State Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No